CLINICAL TRIAL: NCT05931263
Title: A Randomized Controlled Clinical Trial Comparing Chidamide,Carmustine,Etoposide,Cytarabine and Melphalan With BEAM Regimen Combined With Autologus Hematopoietic Stem Cell Transplantation for the Treatment of Newly Diagnosed PTCL
Brief Title: A Randomized Clinical Trial Comparing Chi-BEAM With BEAM Regimen Combined With ASCT for the Treatment of ND PTCL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-T29
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Newly Diagnosed Peripheral T-cell Lymphoma
Keywords: PTCL; Chidemide
MeSH Terms: interventions — BEAM regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-BEAM (Experimental): Chidemide，carmustine, etoposide, cytarabine, and melphalan plus autologous stem cell transplantation
  Interventions: Drug: C-BEAM Regimen
- BEAM (Sham Comparator): carmustine, etoposide, cytarabine, and melphalan plus autologous stem cell transplantation
  Interventions: Drug: BEAM Regimen

INTERVENTIONS:
Drug: C-BEAM Regimen — Chidemide，carmustine, etoposide, cytarabine, and melphalan
  Arms: C-BEAM
Drug: BEAM Regimen — carmustine, etoposide, cytarabine, and melphalan
  Arms: BEAM

SUMMARY:
The goal of this clinical trial is to compare Chi-BEAM With BEAM Regimen Combined With ASCT for the Treatment of ND PTCL.

The main question it aims to answer are:

•Whether Chi-BEAM improves patient survival compared to BEAM group Participants will be given BEAM or Chi-BEAM before ASCT. Researchers will compare the efficacy and safety of the two groups.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled, open trial. The primary endpoint was 2-year PFS The secondary endpoint was： 2-year overall survival (OS). CR rate at 3 months post-transplant evaluation Hematopoietic reconstitution time Non-recurrent mortality (NRM)

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed patients with newly treated PTCL (including NT/ K-cell lymphoma), except for ALK (+), have CR or PR after first-line treatment;
2. Renal function needs to be satisfied: creatinine clearance ≥80ml/min, creatinine less than 160μmol/L; Liver function requirements: ALT and AST≤2 times the upper limit of normal; Total bilirubin ≤2 times the upper limit of normal; Lung function should meet: FEV1, FVC, DLCO≥50% predictive value; Cardiac function must be satisfied: left ventricular ejection fraction ≥50%, asymptomatic arrhythmia.
3. Age between 18 and 65 years old, male and female;
4. ECOG physical strength score 0-1;
5. Neutrophil absolute value ≥1.5×109/L, platelets ≥ 70×109/L, hemoglobin ≥ 90g/L; Number of CD34+ cells ≥ 2.0×106/kg body weight;
6. Expected survival time ≥3 months;
7. Voluntarily sign written informed consent.

Exclusion Criteria:

1. Lymphoma involving the central nervous system
2. Active hepatitis B or C virus infection;
3. Active infection;
4. HIV infected persons;
5. Evidence of cirrhosis or liver fibrosis;
6. Ecg showed QTc > 500ms;
7. Persons with mental disabilities/unable to obtain informed consent;
8. Patients with drug or chronic alcohol abuse that may affect the evaluation of study results;
9. Pregnant and lactating women and women of childbearing age who do not want to take contraceptive measures;
10. The researcher determines that it is not suitable to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
2-y PFS | 2 years
  2-year PFS

SECONDARY OUTCOMES:
2-year OS | 2 years
CR rate at 3 months post-transplant evalutation | 2 years
hematopoietic reconstitution time | 2 years
Non-recurrent mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: wei xu, Principal Investigator — : China, Jiangsu Hematological Department, People's Hospital of Jiangsu Province
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China